CLINICAL TRIAL: NCT02016001
Title: Identification of Effective Fluoride Concentration In Toothpaste For Dental Caries Prevention; A Randomized Controlled Trial
Brief Title: Effective Fluoride Concentration In Toothpaste For Dental Caries Prevention
Acronym: DMFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, DRAEEZA MALIK, dr., Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: draeezamalik; DUHS (Other: DUHS)
Record Dates: First submitted 2013-11-09; First posted 2013-12-19 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Dental Caries
Keywords: fluoride; dental caries; prevention
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- toothpaste 1 (Experimental): tooth paste 1 will be the tested intervention with maximum fluoride concentration (1500ppm), which will be provided to the case group. They will brush the teeth twice daily for 2 minutes
  Interventions: Other: toothpaste 1 with maximum fluoride concentration
- toothpaste 2 (Experimental): toothpaste 2 will be the intervention with 1000 ppm of fluoride, which will be used by control group. They will brush the teeth twice daily for 2 minutes
  Interventions: Other: toothpaste 2 with 1000 ppm of fluoride

INTERVENTIONS:
Other: toothpaste 1 with maximum fluoride concentration — tooth paste 1 will be the tested intervention with maximum fluoride concentration (1500 ppm), which will be provided to the case group. They will brush the teeth twice daily for 2 minutes
  Other Names: locally available tooth paste
  Arms: toothpaste 1
Other: toothpaste 2 with 1000 ppm of fluoride — tooth paste 2 will be the intervention with 1000ppm of fluoride, will be used by the control group. They will brush the teeth twice daily for 2 minutes
  Other Names: locally manufactured toothpaste
  Arms: toothpaste 2

SUMMARY:
to identify the Effective Fluoride Concentration In Toothpaste For Dental Caries Prevention after 18 months of randomized controlled trial.

DETAILED DESCRIPTION:
In developed countries, well-controlled clinical trials have investigated the effective fluoride level in toothpaste and provided irresistible data in relation to the caries controlling efficacy of tooth pastes. But there has been no such data reported in our part of the world. This indicates the need to determine the effective concentration of fluoride in locally manufactured tooth pastes for accomplishment of the goal of prevention against dental caries.

This will be a Parallel Group, Double-Blind, Randomized Controlled Trial, over a period of 18 months. The study will be conducted in a randomly selected school of Karachi city. Participants will be the cohort of regular school children aged 12-14 years. Sample size for the present study attained was 330 (165 in both groups), expected attrition rate will be kept as 15%, so the total sample size is 330 + 50 = 380 (190 in each group).

ELIGIBILITY:
Inclusion Criteria:

1. Regular school children of 12-15 years
2. Presence of at least four molars

Exclusion Criteria:

1. Non- consenting cases
2. Medically/physically compromised children
3. Children under any kind of parallel fluoride regime (systemic or topical)
4. Children consuming diet that is different from routine dietary practices
5. Children using toothpaste with greater than 1100 ppm and less than 500 ppm of fluoride
6. Children found with rampant caries
7. Children found with all filled molars
8. Children with any oral infection abscess, periodontitis etc
9. Dentition with malocclusion
10. Children undergoing orthodontic/prosthodontic treatment
11. Children with Temporo mandibular joint disorder
12. Children who missed the baseline examinations
13. Loss to any follow-up cases

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 380 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
changes in DMFT (decayed, missing filled teeth) scores, over a period of 18 months. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ambrina Qureshi, BDS, M-Phil, Study Director — Head of Community Department, Dow University of Health Sciences, Karachi, Pakistan
Locations (1):
- Shaheen Public School, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Walsh T, Worthington HV, Glenny AM, Appelbe P, Marinho VC, Shi X. Fluoride toothpastes of different concentrations for preventing dental caries in children and adolescents. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD007868. doi: 10.1002/14651858.CD007868.pub2. PMID 20091655
- See also: Walsh T, Worthington HV, Glenny AM, Appelbe P, Marinho VC, Shi X. Fluoride toothpastes of different concentrations for preventing dental caries in children and adolescents. Cochrane Database Syst Rev. 2010;1. — http://www.ncbi.nlm.nih.gov/pubmed/20091655